CLINICAL TRIAL: NCT03671226
Title: Perception of Supportive Care Patients and Caregivers Who Are Seen in the Outpatient Supportive/Palliative Care Center Regarding the Preference of Room Setting and Waiting Time
Brief Title: Preference of Room Setting and Waiting Time in Patients With Advanced, Locally Advanced, or Metastatic Cancer and Their Caregivers Who Are Seen in the Outpatient Supportive/Palliative Care Center
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2018-0573; NCI-2018-01877 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2018-0573 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2018-09-12; First posted 2018-09-14 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: Advanced Malignant Neoplasm; Caregiver; Locally Advanced Malignant Neoplasm; Metastatic Malignant Neoplasm
MeSH Terms: conditions — Neoplasm Metastasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Supportive Care (questionnaire) (Experimental): Patients and their caregivers complete a questionnaire over 15 minutes either in person or over the phone within 3 days after their supportive care center visit.
  Interventions: Other: Questionnaire Administration

INTERVENTIONS:
Other: Questionnaire Administration — Given questionnaire

SUMMARY:
This trial studies the preference of room setting and waiting time in patients with cancer that has spread to nearby tissue or lymph nodes or other places in the body and their caregivers who are seen in the outpatient supportive/palliative care center. Room setting preferences of patients and caregivers may help to understand their opinion regarding direct rooming system in the outpatient supportive/palliative care center.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine patients and caregivers preferences regarding the rooming process in outpatient supportive palliative care clinic, measured by the preference to exam room versus waiting area.

SECONDARY OBJECTIVES:

I. Patients and caregiver perceptions regarding room setting and waiting time in the outpatient supportive care clinic.

II. Extent/experience of team contact in the outpatient supportive care clinic. III. The factors associated with rooming preferences such as age, gender, symptom distress and performance status.

IV. The association between level of distress (physical, psychological, and spiritual distress as measured by Edmonton Symptom Assessment Scale (ESAS) and perception of usefulness of the visit to palliative care center.

V. The attitudes and beliefs toward usefulness of referral to outpatient palliative care.

VI. The correlation between the patient and caregivers preferences.

OUTLINE:

Patients and their caregivers complete a questionnaire over 15 minutes either in person or over the phone within 3 days after their supportive care center visit.

ELIGIBILITY:
Inclusion Criteria:

* Patient: Have advanced cancer, defined as locally advanced, metastatic or incurable disease.
* Patient: Seen at University of Texas M. D. Anderson Cancer Center (UTMDACC) outpatient Supportive Care Center for consultation (first visit).
* Patient: Provided informed consent.
* Patient: Can read and speak English or Spanish.
* Patient: Has a consenting caregiver at the time of the Supportive Care consultation visit.
* Caregiver: Provided informed consent.
* Caregiver: Can read and speak English or Spanish.
* Caregiver: Must be with consenting patient at the time of the Supportive Care consultation visit.

Exclusion Criteria:

* Patient: Delirium diagnosed by palliative care physician or nurse and/or Memorial Delirium Assessment Scale (MDAS) >= 7 or dementia.
* Patient: Inability to read and speak English or Spanish.
* Patient: No caregiver at the time of Supportive Care consultation visit.
* Caregiver: Inability to read and speak English or Spanish.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 406 (Actual)
Dates: Start 2018-09-28 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Preference of exam room over waiting room as soon as checking in until the nurse is ready for a patient assessed using questionnaire | Up to 3 days after visit
  Two sample t-test or Wilcoxon rank sum test, whichever more appropriate, will be used to compare continuous variables of interest between the preference of exam room over waiting area. Chi-squared test or Fisher's exact test, whichever appropriate, will be used to test for associations between each of categorical variables and preference of exam room over waiting area. Univariate/multicovariate logistic regression analysis will be used to explore the demographics and clinical factors associated with rooming preferences.

CONTACTS AND LOCATIONS:
Overall Officials: MarieBerta Vidal, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org